CLINICAL TRIAL: NCT05463198
Title: Evaluation of Physiological Variables and Detection of Blood Loss Using the Zynex Fluid Monitoring System, Model CM-1600
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zynex Monitoring Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZMS-1600-Blood Loss Detection
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Fluid Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Blood Loss (Experimental)
  Interventions: Device: CM-1600

INTERVENTIONS:
Device: CM-1600 — Subjects undergoing blood donation will be connected to the CM-1600 device.

SUMMARY:
The study is a prospective, non-randomized, non-blinded, non-significant risk, multi-center study enrolling up to 500 healthy adult subjects consented to undergo a whole blood donation procedure. The study will involve enrolling subjects that will undergo blood donation wearing the study device (CM-1600 Device) and capture study-required physiological parameters pre-, during, and post-donation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written consent
* Ability and willingness to comply with the study procedures and duration requirements
* 18 years of age or older
* Consented and eligible to undergo a single unit whole blood donation

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Undergone an amputation of any upper extremity
* Diagnosed with dextrocardia
* Subjects who have a pacemaker
* Subjects with body hair density which prevents adequate application of device electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Vitalant Research Institute, Denver, Colorado
  - SunCoast Blood Centers, Bradenton, Florida
  - ClinCept, LLC, Columbus, Georgia
  - Blood Assurance, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.zynexmonitoring.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blood Loss
Started | 351
Completed | 314
Not Completed | 37
Not completed — Withdrawal by Subject | 19
Not completed — Procedure Notes Missing | 18

BASELINE CHARACTERISTICS:
Arm/Group | Blood Loss
Number analyzed (Participants) | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (21.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193
  Male | 121
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 314

OUTCOME MEASURES:

1. Primary Outcome: Change in the Relative Index (RI) After Minor Blood Loss (e.g., 500mL)
Description: The objective of this study is to determine if manual blood loss of up to 500mL of blood can be identified using the non-invasive Zynex CM-1600. This will be measured by determining the percent change in Relative Index (RI) before and after the Blood Draw. The RI is an investigational value which utilizes proprietary algorithms to combine the changes of multiple measured parameters (utilizing a weighted summation of percent change values) which are indicative of relative changes in fluid volume in adult patients into a single value. The RI is a unitless value with no set minimum or maximum, where 100 is a patient's baseline. Based on the nature of the RI itself, a direct interpretation of a positive or negative outcome cannot be derived from the absolute value, instead it could be used to monitor trending of a patient's parameters relative to their baseline.
Time Frame: Recovery period following donation (10 minutes)
Population: 18 subjects were unevaluable; 19 subjects were withdrawn
Measure: Mean (Standard Deviation); unit: Percent change in RI
Arm/Group | Blood Loss
Number analyzed (Participants) | 314
Percent change in RI | 2.9 (151.1)

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded during subject participation and for 24hrs after participation was complete, a total of up to 27hrs.
Arm/Group | Blood Loss
All-Cause Mortality (participants affected / at risk) | 0/351
Serious Adverse Events (participants affected / at risk) | 0/351
Other Adverse Events (participants affected / at risk) | 4/351
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blood Loss (N=351)
Light-headedness due to blood donation procedure (General disorders) | 4 (4) — Subject experienced light-headedness accompanied with nausea or dizziness in response to the blood donation procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT05463198/Prot_SAP_000.pdf